CLINICAL TRIAL: NCT00868361
Title: A Phase 1 Open-label Mass Balance Study to Investigate the Absorption, Metabolism and Excretion of [14C]-Talampanel Following Oral Administration to Healthy Male
Brief Title: A Study to Investigate the Absorption, Metabolism and Excretion of Talampanel
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor recruitment of fast and slow acetylators
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Siyu Liu, M.D., Ph.D., Vice President, Innovative Research and Development and Head of Global Clinical Operations
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAL-MB-100
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Mass Balance; Talampanel; Pharmacokinetics; Metabolism; Metabolites; Healthy Volunteers
MeSH Terms: interventions — talampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Slow and rapid N-acetyl transferase genotypes (Experimental)
  Interventions: Drug: Talampanel (non-radiolabeled), [14C] Talampanel

INTERVENTIONS:
Drug: Talampanel (non-radiolabeled), [14C] Talampanel — 50 mg capsule single dose
  Other Names: TV-7600

SUMMARY:
The purpose of this study is to characterize the chemical breakdown and excretion of talampanel and its break down products in plasma, feces, and urine of healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Males, between 18 and 55 years of age, inclusive
* Body Mass Index range 18.0 to 30.0 kg/m2, inclusive
* Have NAT2 slow or rapid acetylator genotype
* In good health as determined by the investigator
* Negative test for selected drugs of abuse at screening
* Negative screens for Hepatitis B, Hepatitis C and HIV
* Sterile or agrees to use an approved method of contraception from Check-in until 45 days following Clinic Discharge
* Able to comprehend and willing to sign an Informed Consent Form
* Have 1 to 2 bowel movements per day

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, skin, liver, kidney, blood, heart or blood vessel, digestive system, brain or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of stomach or intestinal surgery or resection
* History or presence of an abnormal ECG,
* History of clinically significant alcohol or drug use within 1 year prior to Check-in
* Participation in more than 1 other radiolabeled investigational study drug trial within 12 months prior to Check-in
* Exposure to significant radiation within 12 months prior to Check-in -Use of any tobacco- or nicotine-containing within 6 months prior to Check- in
* Use of any drugs which may interact with the study drug within 30 days prior to Check-in
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 30 days prior to Check-in
* Use of any prescription medications/products within 14 days prior to Check in
* Use of any over-the-counter, non-prescription drugs within 7 days prior to Check-in
* Use of grapefruit or grapefruit-containing foods or beverages within 7 days prior to Check-in
* Use of alcohol- or caffeine-containing foods or beverages within 72 hours prior to Check-in
* Donation of blood from 30 days prior to Screening through Study Completion, inclusive, or of plasma from 2 weeks prior to Screening through Study Completion
* Receipt of blood products within 2 months prior to Check-in
* Any acute or chronic condition that would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To determine the mass balance of [14C]-talampanel. To characterize the metabolism of [14C] talampanel in plasma, feces, and urine. To assess the pharmacokinetics (PK) of total radioactivity, talampanel, and N-acetyl talampanel. | 6-9 days

SECONDARY OUTCOMES:
To explore the effect of N-acetyltransferase 2 (NAT2) genotype on the PK and metabolism of [14C] talampanel. To further assess the safety and tolerability of talampanel. | 6-9 days

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas M Siebers, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Pharmacology Inc., Madison, Wisconsin, United States